CLINICAL TRIAL: NCT03999281
Title: Retrospective Clinical Trial Study of 188 Consecutive Patients to Examine the Effectiveness of a Biological Active Cryopreserved Human Skin Allograft on the Treatment of Diabetic Foot Ulcers and Venous Leg Ulcers
Brief Title: Clinical Trial to Examine Effectiveness of a Human Allograft for Treatment of DFU and VLU
Status: Completed | Type: Observational
Sponsor: Solsys Medical LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SolubleS
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Determine Effectiveness of Theraskin in the Treatment of DFU and VLU

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Foot Ulcers (DFU): Study began with 214 consecutive patient; After excluding patients who did not meet the study criteria, the final eligible cohort consisted of 188 subjects, with 54 with diabetic foot ulcers
  Interventions: Other: Human Allograft (Theraskin)
- Venous Leg Ulcer (VLU): Study began with 214 consecutive patient; After excluding patients who did not meet the study criteria, the final eligible cohort consisted of 188 subjects, with 134 venous leg ulcers.
  Interventions: Other: Human Allograft (Theraskin)

INTERVENTIONS:
Other: Human Allograft (Theraskin) — Biologically active cryopreserved human skin allograft (Theraskin) was used on both cohorts, both diabetic foot ulcer and venous leg ulcer.

SUMMARY:
Retrospective clinical study of 188 patients to examine effectiveness of human cryopreserved allograft in the treatment of diabetic foot ulcers and venous leg ulcers

DETAILED DESCRIPTION:
Retrospective Observational study of 188 consecutive patients to examine the efficacy of biologically active cryopreserved human skin allograft (Theraskin) on the treatment of diabetic foot ulcers and venous leg ulcers

ELIGIBILITY:
Inclusion Criteria:

1. Theraskin applied to lower extremity wound during the study period.
2. Over 18 years of age.
3. Males and Females.
4. lower Extremity wound due to diabetic neuropathy or venous insufficiency.
5. Documented palpable pedal pulse (dorsalis pedis and/or posterior tibialis arteries and/or palpable bypass graft), or ankle brachial index (ABI) in the range of > 0.8 to < 1.1 or Tcpo2 > 40 mm Hg from the foot at the time of the initial allograft applicaton
6. In subjects with multiple wounds only the largest wound receiving the allograft was included and considered the target wound
7. Initial wound size >1 cm 2
8. All wound locations within the lower extremity (defined as below the knee) and wound durations included
9. Concomitant Negative pressure wound therapy was allowed as this could have been an anchoring technique for the allograft
10. Concomitant antibiotics ( topical, oral, or intravenous) were allowed as it was not possible to determine whether administration of antibiotics was due to a true infection at the target wound site.

Exclusion Criteria:

1. Wound etiologies other than diabetic neuropathy or nevous such as trauma, burns, sickle cell anemia, necrobiosis lipoidica , pyoderma gangrenosum.
2. Wound not present for at least 30 days and showing lack of progression for at least 30 days prior to application of Theraskin.
3. Other ulcer treatments besides study allograft during the study period ( study period definition: time of first allograft application up to 20 weeks) were not included in this study. These concomitant treatments specifically include hyperbaric oxygen treatments, venous ablation procedures, revascularization procedures including lower extremity bypass grafts or angioplasties or stents, application of additional growth factors, biologic products containing cells or other tissue-derived products, matrix components, or enzymatic debriders. Subjects were allowed to receive standard of care therapy with the study allograft, which included debridement, moist dressings or compression dressings depending on wound etiology, and off-weighting depending on wound location.
4. Patients with revascularization procedures (defined as lower extremity bypass grafts, angioplasties, or stents) within 30 days of initial TheraSkin application were excluded
5. Patients with successful surgical correction or intervention aimed at improving venous return in the target limb, such as venous ablation procedures, within 30 days of initial TheraSkin application were excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population included ages 18- any age, males 50.5 % and females 49.5%, There was more males in the diabetic subset and more females in the venous subset.
  Percentage by Race: White: 72.3, Black: 17.6, Hispanic: 4.8 and unknown: 5.3
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2003-03-20 (Actual); Primary Completion 2009-09-20 (Actual); Study Completion 2009-09-20 (Actual)

PRIMARY OUTCOMES:
Primary aim was to determine effectiveness of Theraskin together with standard of care | 12-20 weeks
  Theraskin used together with standard of care in healing DFU and VLU wounds

SECONDARY OUTCOMES:
Measure of effectiveness based on healing | 12-20 weeks
  Effectiveness was measured based on the proportion of complete wound closures at 12 and 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Fairfax, Virginia, United States